CLINICAL TRIAL: NCT05977023
Title: NMDA Receptor Modulation for the Treatment of Cognitive Impairment and Perceived Stress in Bipolar I Disorder
Brief Title: NMDA Receptor Modulation for the Treatment of Bipolar I Disorder
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Collaborators: National Science and Technology Council (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CMUH111-REC2-222
Record Dates: First submitted 2023-07-28; First posted 2023-08-04 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Bipolar I Disorder
Keywords: Bipolar I disorder; Bipolar depression; NMDA
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NMDAE (Experimental): An NMDA enhancer
  Interventions: Drug: NMDAE
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo Cap

INTERVENTIONS:
Drug: NMDAE — Use of an NMDA enhancer for the treatment of bipolar depression
  Arms: NMDAE
Drug: Placebo Cap — Use of placebo as a comparator.
  Arms: Placebo

SUMMARY:
At present, the treatment of Bipolar I disorder (BD-I), especially its depressive episode (bipolar depression), is still limited, because there is no effective treatment for the associated cognitive impairment and perceived stress. NMDA receptor (NMDAR) dysfunction is associated with BD-I, particularly its cognitive impairment and perceived stress. This study aims to examine the efficacy and safety of an NMDA enhancer (NMDAE) in the treatment of cognitive impairment and perceived stress in the patients with bipolar depression.

DETAILED DESCRIPTION:
Bipolar I disorder (BD-I) is a severe brain disorder. At present, the treatment of BD-I, especially its depressive episode (bipolar depression), is still limited, because there is no effective treatment for the associated cognitive impairment and perceived stress. This study aims to examine the efficacy and safety of an NMDA enhancer (NMDAE) in the treatment of cognitive impairment and perceived stress in the patients with bipolar depression.

The subjects are bipolar depression patients. They have been treated for bipolar depression for at least four weeks but remain depressive. Participating in this study, they will continue the original treatment, and will be randomized, double-blindly to receive the NMDAE or placebo for 8 weeks. We will measure 6 cognitive domains (including 9 cognitive tests) and quality of life at weeks 0 and 8; and assess the Perceived Stress Scale, Global Assessment of Function (GAF), various scales for clinical symptoms, and side effects at weeks 0, 2, 4, 6, and 8.

The efficacies of NMDAE and placebo will be compared. Chi-square (or Fisher's exact test) will be used to compare differences of categorical variables and t-test (or Mann-Whitney test if the distribution is not normal) for continuous variables between treatment groups. Mean changes from baseline in repeated-measure assessments will be assessed using the generalized estimating equation (GEE). All p values for clinical measures will be based on two-tailed tests with a significance level of 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Are 18 to 65 years of age;
* Satisfy a DSM-5-TR (American Psychiatric Association) diagnosis of BD-I, current episode depressed, after treatment of stable (i.e., at least 4 weeks) and adequate treatment of antipsychotic (quetiapine or lurasidone) and/or mood stabilizer;
* Have a 17-item Hamilton Depression Rating Scale (HAMD) score ≥18 and a Young Mania Rating Scale (YMRS) score ≤7 at baseline;
* Agree to participate in the study and provide informed consent

Exclusion Criteria:

* Current substance abuse or history of substance dependence in the past 6 months
* History of epilepsy, head trauma, stroke or other serious medical or neurological illness which may interfere with the study
* Schizophrenia or other psychotic disorder
* Moderate-severe suicidal risks
* Severe cognitive impairment
* Clinically significant laboratory screening tests (including blood routine, biochemical tests)
* Pregnancy or lactation;
* Inability to follow protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-10-04 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change in Visual Continuous Performance Test | week 0, 8
  Assessment of sustained attention
Change in Wisconsin Card Sorting Test | week 0, 8
  Assessment of abstract and shift set
Change in Logical Memory Test of the Wechsler Memory Scale | week 0, 8
  Assessment of episodic memory
Digit Span | week 0, 8
  Assessment of verbal working memory
Spatial Span | week 0, 8
  Assessment of nonverbal working memory
Category Fluency | week 0, 8
  Assessment of speed of processing
Trail Marking A | week 0, 8
  Assessment of speed of processing
WAIS-III Digit Symbol-Coding | week 0, 8
  Assessment of speed of processing
Mayer-Salovey-Caruso Emotional Intelligence Test (MSCEIT) V2.0 | week 0, 8
  Assessment of social cognition
Change in Perceived Stress Scale in Perceived Stress Scale | week 0, 2, 4, 6, 8
  Assessment of stress and anxiety symptoms Minimum value: 0, maximum value:56, the higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Change in Quality of life (SF-36) | week 0, 8
Change in Global Assessmeint of Functioning | Week 0, 2, 4, 6, 8
  Assessment of global improvement. Minimum value: 1, maximum value:100, the higher scores mean a better outcome.
Change in Hamilton Rating Scale for Depression | Week 0, 2, 4, 6, 8
  Assessment of depressive symptoms. Minimum value: 0, maximum value:52, the higher scores mean a worse outcome.
Change in Montgomery-Åsberg Depression Rating Scale | Week 0, 2, 4, 6, 8
  Assessment of depressive symptoms. Minimum value: 0, maximum value:60, the higher scores mean a worse outcome.
Change in Young Mania Rating Scale | Week 0, 2, 4, 6, 8
  Assessment of manic symptoms. Minimum value: 0, maximum value:60, the higher scores mean a worse outcome.
Change in Beck Scale for Suicide Ideation | Week 0, 2, 4, 6, 8
  Assessment of Suicide Ideation. Minimum value: 0, maximum value:38, the higher scores mean a greater risk of suicide.
Change in Clinical Global Impression Scale | Week 0, 2, 4, 6, 8

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychiatry, China Medical University Hospital, Taichung, Taiwan